CLINICAL TRIAL: NCT05177419
Title: Effects of Lysergic Acid Diethylamide (LSD) on Neuroplasticity in Healthy Human Subjects
Brief Title: Effects of LSD on Neuroplasticity in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Fribourg (Other)
Responsible Party: Principal Investigator, Gregor Hasler, Professor, University of Fribourg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LSD-Plasticity
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose LSD (Experimental): High dose of lysergic acid diethylamide
  Interventions: Drug: Lysergic Acid Diethylamide
- Low-dose LSD (Active Comparator): Low dose of lysergic acid diethylamide
  Interventions: Drug: Lysergic Acid Diethylamide

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide — 100 micrograms LSD base
  Other Names: LSD
  Arms: High-dose LSD
Drug: Lysergic Acid Diethylamide — Low dose of LSD base
  Other Names: LSD
  Arms: Low-dose LSD

SUMMARY:
Neuroplasticity is the brain's ability to reorganize itself and adapt in response to changing environmental conditions or pathological stimuli. LSD is a potent psychedelic drug which has been able to rapidly stimulate neuroplasticity in animal studies. Various authors have speculated that changes in neuroplasticity may contribute to LSD's long-term effects, but there is still little direct evidence that LSD or other psychedelics enhance neuroplasticity in humans. The goal of this study is to investigate the effects of LSD on several measures of neuroplasticity in healthy human subjects.

DETAILED DESCRIPTION:
Neuroplasticity is the brain's ability to reorganize itself and adapt in response to changing environmental conditions or pathological stimuli. Its dysregulation may play a role in the etiology of depression and anxiety disorders, and it is also essential for recovery from neural injury and stroke.

LSD is a potent psychedelic drug and a member of the psychoplastogen family of small molecules, which are able to rapidly stimulate neuroplasticity in cortical neurons following a single dose. Previous research suggests that changes in neuroplasticity may contribute to LSD's long-term effects, which include increases in subjective well-being and life satisfaction, reduced anxiety, and increased openness to experience. Additionally, there is some evidence that LSD and other psychedelics could be viable clinical treatments for depression, anxiety, and addictive disorders, and that changes in neuroplasticity may underlie this clinical potential. However, there is still little direct evidence that LSD or other psychoplastogens enhance cortical plasticity in humans.

The goal of this study is to investigate the effects of LSD on several measures of neuroplasticity in healthy human subjects, as well as other abilities and traits thought to be related to neuroplasticity. Determining whether LSD enhances cortical plasticity, how long this may last, where in the brain it occurs, and what it means for cognition and emotion is essential for understanding LSD's long-term effects, including but not limited to its clinical potential.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-55
2. Body mass index 18-29
3. Right-handed as assessed by the Edinburgh Handedness Inventory (score > 60)
4. Fluent understanding of German
5. Willingness to adhere to study protocol
6. Willingness to refrain from taking illicit psychoactive substances for the duration of the study
7. Willingness to refrain from consuming alcohol for 24 hours before each study appointment.
8. Willingness to not operate a motor vehicle or other heavy machinery 48 hours after each substance administration.
9. Women of childbearing potential must be willing to use effective birth control during the study (e.g. birth control pill; condoms must be combined with a second reliable method).
10. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests will be repeated before each treatment day and must remain negative.
11. A friend or relative must be available to accompany the participant home following LSD appointments.

Exclusion Criteria:

1. Severe chronic or acute medical condition
2. History of any seizure disorder, stroke, or cardiovascular illness
3. History of severe head trauma resulting in loss of consciousness
4. Personal or family history (first-degree relative) of psychotic disorders
5. Current or previous major neurological or psychiatric disorder within the last 3 years (e.g. major depression, anorexia, substance use disorder),
6. History of medically relevant suicide attempts
7. Current use of psychoactive medications
8. Lifetime use of hallucinogens, dissociatives, or entheogens more than 10 times, or any time within the previous three months
9. Regular (daily or near-daily) use of cannabis, alcohol, nicotine, or illicit substances
10. Pregnant or nursing women
11. Presence of any implanted, metal or electronic devices (e.g. pacemaker)
12. Recent or current participation in another clinical trial

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Change in motor evoked potential amplitude after paired associative stimulation (PAS) | Baseline, 8 hours post-treatment, 1 day post-treatment, 1 week post-treatment
  Assessment of capacity for neuroplastic changes in the motor cortex

SECONDARY OUTCOMES:
Change in auditory event-related potential (ERP) amplitude after tetanic stimulation | Baseline, 8 hours post-treatment, 1 day post-treatment, 1 week post-treatment
  Assessment of capacity for neuroplastic changes in the auditory cortex
Plasma and serum levels of brain-derived neurotrophic factor (BDNF) | Baseline, 8 hours post-treatment, 1 day post-treatment, 1 week post-treatment
  Marker of neuroplasticity
Motor learning ability | 1 day post-treatment
  Speed and accuracy on a motor learning task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Fribourg, Fribourg, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided